CLINICAL TRIAL: NCT05480722
Title: Central Sodium Sensing: Implications for Blood Pressure Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, William Farquhar, Professor, University of Delaware
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1808532
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Salt Sensitivity of Blood Pressure
MeSH Terms: interventions — Saline Solution, Hypertonic; Furosemide

STUDY DESIGN:
Intervention Model Description: single blinded crossover design
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hypernatremia + Furosemide first, then Hypernatremia without Furosemide (Experimental): Participants in this arm will undergo blood-oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) on two separate days. On the first testing day, participants will receive a hypertonic saline infusion with NKCC2 antagonism (furosemide). On the second testing day, participants will receive a hypertonic saline infusion without NKCC2 antagonism (furosemide). This will enable us to examine sodium sensing mechanisms. The two conditions will be separated by at least 1 week washout. The hypertonic saline will be a 3% NaCl solution infused intravenously at a rate of 0.15 ml/kg/min for 30 minutes; the furosemide will be infused intravenously as a 40 mg bolus in 4mL of isotonic saline (0.9% NaCl) immediately prior to the hypertonic saline infusion.
  Interventions: Other: Hypertonic Saline with furosemide; Other: Hypertonic Saline without furosemide
- Hypernatremia without Furosemide first, then Hypernatremia + Furosemide (Experimental): Participants in this arm will undergo blood-oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) on two separate days. On the first testing day, participants will receive a hypertonic saline infusion without NKCC2 antagonism (furosemide). On the second testing day, participants will receive a hypertonic saline infusion with NKCC2 antagonism (furosemide). This will enable us to examine sodium sensing mechanisms. The two conditions will be separated by at least 1 week washout. The hypertonic saline will be a 3% NaCl solution infused intravenously at a rate of 0.15 ml/kg/min for 30 minutes; the furosemide will be infused intravenously as a 40 mg bolus in 4mL of isotonic saline (0.9% NaCl) immediately prior to the hypertonic saline infusion.
  Interventions: Other: Hypertonic Saline with furosemide; Other: Hypertonic Saline without furosemide

INTERVENTIONS:
Other: Hypertonic Saline with furosemide — Subjects will undergo MRI with a hypertonic saline infusion with NKCC2 antagonism (furosemide). The hypertonic saline will be a 3% NaCl solution infused intravenously at a rate of 0.15 ml/kg/min for 30 minutes; the furosemide will be infused intravenously as a 40 mg bolus in 4mL of isotonic saline (0.9% NaCl) immediately prior to the hypertonic saline infusion.
Other: Hypertonic Saline without furosemide — Subjects will undergo MRI with a hypertonic saline infusion. The hypertonic saline will be a 3% NaCl solution infused intravenously at a rate of 0.15 ml/kg/min for 30 minutes.

SUMMARY:
The ability of the brain to sense changing sodium levels in the blood is critical in mediating the neurohumoral responses to hypernatremia, however, the mechanisms underlying sodium sensing in humans is poorly understood. The purpose of this study is to identify key sodium-sensing regions of the human brain in older adults and determine if the Na-K-2Cl co-transporter mediates the neurohumoral response to acute hypernatremia. Completion of this project will increase our understanding of blood pressure regulation, which has major public health implications.

DETAILED DESCRIPTION:
The prevalence of hypertension is very high in older adults, and a major factor in hypertension is salt sensitivity of blood pressure (BP) and elevated sympathetic nerve activity (SNA). However, we know very little about how the human brain 'senses' sodium, and what molecular mechanisms are involved. Rodent studies have identified specialized sodium chloride (NaCl)-sensing neurons in the circumventricular organs (CVOs), which mediate NaCl-induced changes in SNA, arginine vasopressin (AVP), and BP. Recent data suggest the Na-K-2Cl co-transporter (NKCC2) is not kidney specific but is also expressed in brain regions that regulate whole body NaCl and water homeostasis. In addition, NKCC2 is accessible by drugs in the circulation since the CVOs lack a complete blood brain barrier. The objective of this R21 is to identify key NaCl-sensing regions of the brain in older adults and determine if NKCC2 mediates the neurohumoral response to acute hypernatremia. We seek to translate the prior rodent findings to humans by assessing neuronal activation (using blood oxygen level dependent functional magnetic resonance imaging, BOLD fMRI) as well as thirst, AVP, SNA and BP during an acute hypernatremic stimulus, with and without an NKCC2 antagonist (furosemide). This will enable us to assess the role of NKCC2 in NaCl sensing. The overall hypothesis is that acute hypernatremia will elicit detectable changes in the BOLD fMRI signal and increase thirst, AVP, SNA, and BP largely through NKCC2 in healthy older adults. Accordingly, the first specific aim is to identify the areas of the human brain that respond to acute hypernatremia and determine the role of NKCC2 in central NaCl- sensing. Acute hypernatremia will be induced with a 30-minute infusion of 3% NaCl delivered intravenously. Brain activity during the hypertonic saline infusion will be measured in regions such as the organum vasculosum laminae terminalis, subfornical organ, anterior cingulate cortex, hypothalamus, and insular cortex. The second specific aim is to determine the effect of acute hypernatremia on thirst, AVP, SNA, and BP, and determine the role of NKCC2 in mediating these responses. Salt sensitivity of BP will be individually assessed and comparisons will be made between those with a salt resistant and salt sensitive phenotype; we anticipate that acute hypernatremia will elicit changes in the BOLD fMRI signal and SNA & AVP in all subjects, but the responses will be greater in those who are classified as salt sensitive. This would represent the first trial in healthy human subjects to identify a putative brain NaCl-sensing co-transporter, and we think the scope and innovative approaches are ideal for the R21 funding mechanism. Older adults are prone to hypertension, so it is critically important to understand how normotensive older adults centrally sense sodium, to provide a needed foundation for exploring the mechanistic underpinning of salt sensitive hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 45 years
* Blood pressure: >100/60 mmHg and <130/80 mmHg
* BMI: 18.5 kg/m2 - 30 kg/m2
* Serum potassium: 3.5 mmol/L - 5.5 mmol/L

Exclusion Criteria:

* Age: < 18 years or > 45 years
* Blood pressure: < 100/60 mmHg or > 130/80 mmHg
* BMI: < 18.5 kg/m2 or > 30 kg/m2
* Serum potassium: < 3.5 mmol/L or > 5.5 mmol/L
* Abnormal ECG
* History of - cardiovascular, cancer, metabolic, respiratory, renal disease
* Hormone replacement therapy
* Current tobacco or nicotine use
* Pregnant or nursing mothers
* Major brain injury (concussions do not count)
* Clinically diagnosed psychiatric or neurological disorder
* Clinically diagnosed anxiety or depression
* Psychiatric, neurological, anxiety or depression medications
* Hypertension medications
* Sulfonamide drug allergy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Farquhar, PhD, Principal Investigator — University of Delaware
Locations (1):
- William B Farquhar, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately
Access Criteria: Upon reasonable request

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 participants were consented into the study. However, prior to starting an intervention, participants underwent a medical screening to ensure they qualify for the study. During this process, 7 participants failed the screening and 10 participants withdrew by choice. Thus, these 17 participants did not begin an intervention. This is why we only report a total of 12 participants (9+3) enrolled in the participant flow.
Groups:
- Hypernatremia + Furosemide First, Then Hypernatremia Without Furosemide: Participants in this arm underwent blood-oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) on two separate days. On the first testing day, participants received a hypertonic saline infusion with NKCC2 antagonism (furosemide). On the second testing day, participants received a hypertonic saline infusion without NKCC2 antagonism (furosemide).
- Hypernatremia Without Furosemide First, Then Hypernatremia + Furosemide: Participants in this arm underwent blood-oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) on two separate days. On the first testing day, participants received a hypertonic saline infusion without NKCC2 antagonism (furosemide). On the second testing day, participants received a hypertonic saline infusion with NKCC2 antagonism (furosemide).
Period: Overall Study
Arm/Group | Hypernatremia + Furosemide First, Then Hypernatremia Without Furosemide | Hypernatremia Without Furosemide First, Then Hypernatremia + Furosemide
Started | 9 | 3
Completed | 4 | 2
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants who completed the hypertonic saline infusion protocol both with and without NKCC2 antagonism (furosemide). This is combining participants assigned to the Hypernatremia + Furosemide first, then Hypernatremia without Furosemide Arm and the Hypernatremia without Furosemide first, then Hypernatremia + Furosemide Arm.
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity Between the Subfornical Organ and Organum Vasculosum of the Lamina Terminalis (Z-score)
Description: Functional connectivity between sodium sensing circumventricular organs (subfornical organ (SFO) and organum vasculosum of the lamina terminalis(OVLT)) was calculated (expressed as the z-score). Functional connectivity is a measure of the the correlation (or synchronization) of the blood oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) signal time course between two brain regions. Pearson correlations were computed between the BOLD fMRI signal in the SFO and OVLT in a seed-to-seed functional connectivity analysis. Pearson correlations were converted to Z-scores using a Fisher's transform. A Z-score of 0 indicates no correlation between the BOLD fMRI signal between these 2 brain regions; a higher score indicates a greater, positive correlation between the BOLD fMRI signal in these 2 brain regions; a lower score indicates a greater, negative correlation between the fMRI signal in these 2 brain regions. This data does not have any clinical thresholds.
Time Frame: Functional connectivity (FC) was calculated at baseline (~10 min). Then, participants received a 30-minute hypertonic saline infusion (HSI) with or without furosemide before. FC was calculated during the early (0-15 min) and late phase (15-30 min) of HSI.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Hypertonic Saline Infusion Without Furosemide: Data from participants functional magnetic resonance imaging (fMRI) scan at which they received the hypertonic saline infusion without NKCC2 antagonism (furosemide).
- Hypertonic Saline Infusion + Furosemide: Data from participants functional magnetic resonance imaging (fMRI) scan at which they received the hypertonic saline infusion with NKCC2 antagonism (furosemide).
Arm/Group | Hypertonic Saline Infusion Without Furosemide | Hypertonic Saline Infusion + Furosemide
Number analyzed (Participants) | 6 | 6
z-score
  Baseline (Immediately pre-furosemide and/or hypertonic saline infusion) | 0.258490 (0.105129) | 0.359145 (0.268795)
  Early Phase (0-15 minutes of hypertonic saline infusion) | 0.207372 (0.196048) | 0.169055 (0.169819)
  Late Phase (15-30 minutes of hypertonic saline infusion) | 0.272881 (0.130301) | 0.097043 (0.066845)

ADVERSE EVENTS:
Time Frame: From participant's initial enrollment through their study completion, an average of about 3 months for each participant.
Groups:
- Hypernatremia + Furosemide: For this intervention, participants underwent blood-oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) while they received a hypertonic saline infusion with NKCC2 antagonism (furosemide)
- Hypernatremia Without Furosemide: For this intervention, participants underwent blood-oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) while they received a hypertonic saline infusion without NKCC2 antagonism (furosemide).
Arm/Group | Hypernatremia + Furosemide | Hypernatremia Without Furosemide
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
The study is limited by small sample size; the SFO and OVLT are small regions of interest, making accurate identification challenging; and a small number of participants completed the furosemide protocol, due to needing to urinate, making identification of the mechanism of sodium sensing difficult. The diet component of the protocol originally planned was made optional and few completed it due to the challenges of administering furosemide. We were unable to measure plasma vasopressin (AVP).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT05480722/Prot_SAP_000.pdf